CLINICAL TRIAL: NCT04057326
Title: A Randomized, Double-Blind, Placebo-Controlled Multicenter Clinical Study to Evaluate the Safety and Efficacy of Oryz-Aspergillus Enzyme and Pancreatin Tablet in Improving Malnutrition in Patients With Cirrhosis
Brief Title: A Study of Oryz-Aspergillus Enzyme and Pancreatin Tablet in Patients With Cirrhosis and Malnutrition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Kangzhe Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Combizym-PEM-001
Record Dates: First submitted 2019-08-02; First posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Pancreatin; Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oryz-Aspergillus Enzyme and Pancreatin Tablet Arm (Active Comparator): Oryz-Aspergillus Enzyme and Pancreatin Tablet ,2 tablets/time, 3 times daily. Study drug will be administered orally.
  Interventions: Drug: Oryz-Aspergillus Enzyme and Pancreatin Tablet
- Placebo Arm (Placebo Comparator): Placebo,2 tablets/time, 3 timesdaily. Study drug will be administered orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oryz-Aspergillus Enzyme and Pancreatin Tablet — 2 tablets/time, 3 times daily,Oral Administration.
  Other Names: Treatment Group :Combizym
  Arms: Oryz-Aspergillus Enzyme and Pancreatin Tablet Arm
Drug: Placebo — 2 tablets/time, 3 times daily,Oral Administration.
  Other Names: Control Group
  Arms: Placebo Arm

SUMMARY:
The investigation is a randomized, double-blind, placebo involved and multi-center clinical trial. All subjects are assigned to 2 groups, including Oryz-Aspergillus Enzyme and Pancreatin tablet group (treatment group) and the placebo group (control group). Treatment group includes 99 subjects, while control group includes 33 subjects. They receive investigational drug 2 tablets/times, tid, p.o. for 180 days.

DETAILED DESCRIPTION:
* A total of 132 subjects with cirrhosis were divided into 3 subgroups by Child-Pugh score, which were Child-pugh Class A, B, and C, respectively. Each subgroup includes 44 subjects, which were randomly assigned to the Oryz-Aspergillus Enzyme and Pancreatin tablet group (treatment group) and the placebo group (control group) in a ratio of 3: 1 (33: 11).
* Patients who have signed the Informed Consent Form and are eligible for the entry criteria will be randomly assigned to either the Oryz-Aspergillus Enzyme and Pancreatin tablet group or the placebo group. No matter which group the subjects is assigned, he/she would receive treatment drugs through oral administration for 180 days, during which the participant will not take any investigational drug.
* The differences in nutritional status between treatment group and control group will be compared in 90 and 180 days by MAMC and SGA.

ELIGIBILITY:
Inclusion Criteria:

* The age is range from 18 to 70 years old.
* Sex is not limited.
* Confirmed cirrhosis (pathologic or radiological rationale) with a mid-upper arm muscle circumference (MAMC) < 90% of the standard value.
* The subject or his family (guardians) agreed to participate in the study and signed the informed consent form.

Note: MAMC formula: mid-arm muscle circumference (cm) = mid-arm circumference (cm) - 3.14 × triceps skinfoldthickness. Standard values: 25.3 cm for adult males and 23.2 cm for adult females.

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the following criteria:

* Pregnant, lactating women or women who do not exclude the possibility of pregnancy;
* Total serum bilirubin ≥ 5 times the upper limit of normal;
* Serum creatinine ≥ 1.2 times the upper limit of normal;
* Prothrombin time ≥ 18 seconds;
* Those who have an allergy to Oryz-Aspergillus Enzyme and Pancreatin Tablet and their related ingredients;
* Subjects who are not able to eat orally for any reason;
* Subjects with a history of previous intestinal obstruction;
* Subjects with acute abdominal pain within 2 months prior to the start of the study;
* Subjects with electrolyte (sodium, potassium, chlorine) disorders that cannot be corrected prior to the start of the study, if electrolyte (sodium, potassium, chlorine) disorders have occurred, have been corrected and stabilized for more than 1 month prior to the start of the study;
* Subjects with prior hepatic encephalitic stage II or higher;
* History of refractory ascites with moderate or higher ascites within 2 weeks prior to the start of the study;
* Subjects with symptoms of gastrointestinal bleeding such as melena and hematemesis within 2 weeks prior to the start of the study;
* Those who have used antibiotics within 2 weeks prior to the start of the study;
* Subjects who experienced other conditions that could affect the study: Subjects who had acquired or primary, secondary immune system conditions (except primary autoimmune liver disease) such as major cardiopulmonary disease, diabetes mellitus, tumors, HIV infection, and other conditions that required long-term hormonal therapy;
* Substance abuse: Alcohol abuse (80 g/day) for < 6 months with a history of intravenous or/and inhaled drugs (drugs) in the last two years;
* Subjects with chronic viral hepatitis B/C who started and/or adjusted their antiviral regimen within 6 months prior to the start of the study;
* Subjects with a history of surgery within 6 months prior to the start of the study;
* Subjects with autoimmune liver disease who started or adjusted their regimen within 6 months prior to the start of the study (i.e., subjects who have started treatment for the aetiology with no change in treatment regimen and drug dose in the new addition of ursodeoxycholic acid or hormones, immunosuppressants, etc., in June)
* Those who participated in other drug trials within 3 months prior to the start of the study;
* Any subject who is considered by the investigator to be unable to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2019-08-30 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-03-28 (Estimated)

PRIMARY OUTCOMES:
1. Change in nutritional status by Mid-Arm Muscle Circumference (MAMC) evaluation, the unit of MAMC is centimeter(cm). | 180 days
  The change in nutritional status of subjects at 180 days was evaluated by MAMC. MAMC, as a marker of lean muscle mass, is calculated using the standard formula: MAMC = MAC-(3.14 x TSF thickness).
  MAC: mid-arm circumference TSF : triceps skinfold thickness
2. Change in nutritional status by Subjective Global Assessment (SGA) evaluation. | 180 days
  The change in nutritional status of subjects at 180 days was evaluated by SGA Form.
  The nutritional status of the subjects was improved if any of the index reached the "effective" standard.